CLINICAL TRIAL: NCT02173119
Title: Can Quantitative MRI After Conventional Transarterial Chemoembolization (cTACE) Help Predict Survival ?
Brief Title: Can Quantitative MRI After cTACE Help Predict Survival ?
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Guerbet (Industry); Northwestern University (Other)
Responsible Party: Principal Investigator, Sarah B. White, MD, Assistant Professor of Radiology, Medical College of Wisconsin
Other Study IDs: PRO22746
Record Dates: First submitted 2014-06-17; First posted 2014-06-24 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular; Carcinoma; HCC; lipiodol
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCC patients having MRI post-TACE: HCC patients who have undergone conventional lipiodol based chemoembolization.
  Interventions: Other: MRI post-TACE

INTERVENTIONS:
Other: MRI post-TACE — Perform lipiodol delivery measurements with MRI post-TACE.

SUMMARY:
Transcatheter arterial chemoembolization (TACE) is a widely accepted palliative therapy for the treatment of HCC. Palliative means that it does not cure the disease prolongs your life and improves quality of life. During TACE, a mixture of chemotherapy drugs is combined with an oil called lipiodol. Lipiodol has a role as both drug carrier and embolic agent (a material that blocks blood flow to tumors). The lipiodol/chemotherapy mixture is injected into an artery (blood vessel) directly supplying blood to a HCC tumor.

Lipiodol is made up of fat and water which can be seen on MRI. Therefore, MRI can be used to quantify the amount of lipiodol delivered to the HCC tumors.

In this study, the investigators want to see if patient survival is related to the amount of lipiodol delivered to HCC tumors.

ELIGIBILITY:
Inclusion Criteria:

* Prospective studies will be performed in 20 patients with Hepatocellular Carcinoma (HCC) independently scheduled to undergo TACE; tumors in each of these candidates will already have been deemed un-resectable.
* Reasons may include

  * concurrent co-morbidities including cardiac or respiratory compromise
  * recurrent or multi-lobar disease
  * cirrhosis or portal hypertension
  * vascular invasion
  * high tumor burden
  * contraindications to general anesthesia.
* Diagnosis of HCC will have been established by a) biopsy or b) non-invasively, based upon > 2cm diameter tumor with characteristic imaging findings in the setting of cirrhosis.
* Male or female aged 18 to 89 years, all ethnicities

Exclusion Criteria:

* Infiltrative or diffuse HCC.
* Does not meet inclusion criteria.
* Pregnant women.
* Individuals with pacemakers or other non-MRI compatible metallic implants.
* Hemodialysis patients or patients with severely impaired renal function.
* Individuals with severe claustrophobia or unwilling to get a MRI.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma (HCC or cancer of the liver) and will soon undergo one or more transcatheter arterial chemoembolization (TACE) procedure(s).
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-08; Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Imaging response | Every 4-6 weeks during active treatment and then every 3-6 months, up to 5 years or death.
  Imaging response will be assessed according to 3D European Association for the Study of the Liver (EASL) criteria. EASL criteria propose using contrast enhanced (CE) images to measure viable volumes. We will transfer all images to a computer workstation. We will measure 'viable' enhancing tumor volumes at each interval and percent change in viable tumor volume (change from baseline). We will correlate lipiodol delivery measurements to primary outcomes post-therapy.

SECONDARY OUTCOMES:
Clinical response | Every 4-6 weeks during active treatment and then every 3-6 months, up to 5 years or death.
  Clinical response will be measured using Eastern Cooperative Oncology Group (ECOG) performance status classification. We will consider a change of 0.5 ECOG levels to be clinically significant.
Adverse Events | Every 4-6 weeks during active treatment and then every 3-6 months, up to 5 years or death.
  Adverse Events will be measured according to the Common Terminology Criteria (NCI CTC) version 3.0 criteria for each patient. We will define Grades 0-2 as tolerance to therapy and Grades 3 or 4 as toxic.
Time-to-Tumor Progression | Every 4-6 weeks during active treatment and then every 3-6 months, up to 5 years or death.
  Time-to-tumor progression will be assessed by monitoring viable tumor volumes post-TACE and defining progression as a >44% volume increase (3D EASL criteria).
Survival | Every 4-6 weeks during active treatment and then every 3-6 months, up to 5 years or death.
  We will determine the number of days from first treatment to last follow-up to calculate the median days of overall survival after first treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah B. White, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin/Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gordon AC, Lewandowski RJ, Li W, Zhong X, Kannengiesser SAR, Miller FH, Salem R, Rilling WS, Larson AC, White SB. Chemical Shift MRI Monitoring of Chemoembolization Delivery for Hepatocellular Carcinoma: Multicenter Feasibility of Initial Clinical Translation. Radiol Imaging Cancer. 2023 May;5(3):e220019. doi: 10.1148/rycan.220019. PMID 37233207